CLINICAL TRIAL: NCT04562922
Title: LIFEMEL Efficacy in Preventing Haematopoietic Toxicity in Patients Treated With Chemotherapy
Acronym: LEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VitalMel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LEO
Record Dates: First submitted 2020-08-27; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Neutropenia; Adverse Event
MeSH Terms: conditions — Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifemel (Experimental): LifeMel is bee-honey obtained using Zuf Globus Ltd technology: it is produced in Israel and distributed by VitalMel in Italy. In Italy Ministry of Health has listed it as a food supplement.
  Two tea spoons (5 g each) of honey were administered to subjects on each day of the chemotherapy treatment.
  Interventions: Dietary Supplement: Lifemel

INTERVENTIONS:
Dietary Supplement: Lifemel

SUMMARY:
LEO trial was designed to assess the benefit of administering LifeMel to prevent myelotoxicity in patients affected by solid neoplasm undergoing antiblastic chemotherapy treatment at low to moderate risk of febrile neutropenia. Secondary endpoints of LEO trial were assessing impact of LifeMel in preventing anaemia and thrombocytopenia.

DETAILED DESCRIPTION:
The LEO trial was designed to assess the benefit of administering LifeMel, a honey from bees obtained using Zuf Globus Ltd technology, produced in Israel and listed by the Ministry of Health in Italy as a food supplement. This study aims to highlight a possible role of Lifemel in preventing neutropenic events, as well as reducing anaemia and thrombocytopenia following the administration of chemotherapy in patients with a histological or clinical diagnosis of solid neoplasia undergoing first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 years old
* histological or clinical diagnosis of solid neoplasia
* indication for chemotherapy treatment with regimens at moderate risk of neutropenia fever - duration of chemotherapy treatment more than 3 months

Exclusion Criteria:

* known intolerances to honey containing compounds
* decompensated diabetes or severe glucose intolerance
* diseases or therapies significantly affecting the neutrophil count
* concurrent use of G-CSF as primary or secondary prophylaxis in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2014-05-26 (Actual); Study Completion 2016-04-04 (Actual)

PRIMARY OUTCOMES:
Neutropenia | Three months for each patient
  Neutrophil count has been measured the same day or the day before starting every chemotherapy cycle and at expected nadir (between the 7th and 12th day after chemotherapy) in the first 3 months.
  A patient was considered 'responder' if no episodes of neutropenia was observed during first 3 months of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pietro Sponghini, Principal Investigator — Department of Oncology, A.O.U. Maggiore della Carità, Novara, Italy.

REFERENCES:
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Abdel-Razeq H, Hashem H. Recent update in the pathogenesis and treatment of chemotherapy and cancer induced anemia. Crit Rev Oncol Hematol. 2020 Jan;145:102837. doi: 10.1016/j.critrevonc.2019.102837. Epub 2019 Nov 26. PMID 31830663
- [Background] Zidan J, Shetver L, Gershuny A, Abzah A, Tamam S, Stein M, Friedman E. Prevention of chemotherapy-induced neutropenia by special honey intake. Med Oncol. 2006;23(4):549-52. doi: 10.1385/MO:23:4:549. PMID 17303914